CLINICAL TRIAL: NCT07388134
Title: Effects of Virtual Reality Based High-intensity Interval Training in Chronic Low Back Pain
Brief Title: Virtual Reality Based High-intensity Interval Training in Chronic Low Back Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, Irene Torres Sánchez, PhD, Universidad de Granada
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HIIT_DLC
Record Dates: First submitted 2026-01-23; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Chronic Low-back Pain (cLBP)
MeSH Terms: interventions — Population Groups; High-Intensity Interval Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual reality-based high intensity interval training (VR-HIIT) group (Experimental)
  Interventions: Other: Virtual reality based high intensity interval training (VR-HIIT) group
- High intensity interval training (HIIT) group (Active Comparator)
  Interventions: Other: High intensity interval training (HIIT) group

INTERVENTIONS:
Other: Virtual reality based high intensity interval training (VR-HIIT) group — A single session of 70-90 minutes.
  * Pain neuroscience education
  * VR-HIIT. HIIT session will follow the outline: warm-up and HIIT. VR component will be carried out with the Nintendo Switch.
  Arms: Virtual reality-based high intensity interval training (VR-HIIT) group
Other: High intensity interval training (HIIT) group — A single session of 70-90 minutes.
  * Pain neuroscience education
  * HIIT. HIIT session will follow the outline: warm-up and HIIT.
  Arms: High intensity interval training (HIIT) group

SUMMARY:
One of the most prevalent causes of pain on a global scale is chronic musculoskeletal pain. Low back pain is a prevalent manifestation of chronic musculoskeletal pain.

There are a wide vary of no pharmacologic treatment for chronic pain. From a physiotherapy perspective, the chronic pain management should be oriented towards increasing the self-management of people with chronic pain. The management components in question are therapeutic exercise and education.

High-intensity interval training (HIIT) is a novel therapeutic exercise strategy that has been shown to reduce pain and disability in chronic low back pain. It is a hopeful strategy to enhance motivation to treatment. Pain neuroscience education (PNE) has also been demonstrated to enhance pain and disability in chronic low back pain. Finally, virtual reality (VR) has been demonstrated to be effective in the chronic low back pain management.

Despite the benefits mentioned in these three therapies being isolated, there are no studies that have compared VR-based HIIT (VR-HIIT) with PNE in chronic low back pain. The use of these interventions may increase the intervention benefits. The investigators hypothesise that VR-HIIT with PNE can reduce pain intensity, enhance fear of movement and improve motivation for treatment in chronic low back pain. Therefore, the aim of this study is to evaluate the effects of VR-HIIT with PNE in chronic low back pain.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18-65 years
* Chronic low back pain
* Pain intensity ≥ 3 points with the numeric pain rating scale
* Ability to walk ≥ 15 minutes
* Wish to participate in the study and sign the informed consent

Exclusion Criteria:

* Pregnancy
* Patients with severe comorbidities that interfere with the ability to perform the study
* People who are currently participating in another study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2026-02-09 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | Baseline, during the intervention and 48-72h post-intervention
  To assess pain intensity using the Numeric Pain Rating Scale. Scores range from 0 (no pain) to 10 (worst pain imaginable). Higher scores indicate greater intensity.
Pain pressure threshold | Baseline and 48-72h post-intervention
  To assess pain pressure threshold. The measurement will be taken in the paravertebral and tibialis anterior muscles with the algometer Force One FPIX 50. The measurement points will be lumbar region bilaterally 5 cm from the spinous processes of L3 and L5; and right tibialis anterior, 5 cm below the tibial tuberosity. The assessor will place the algometer perpendicular and applied increasing pressure. until the pressure became painful. The mean of 3 measurements was recorded.
Pain modulation | Baseline and 48-72h post-intervention
  To assess pain modulation using algometer Force One FPIX 50. The pressure pain threshold will be evaluated in the tibialis anterior muscle and the deltoid muscle. Then the conditioning stimulus will be introduced. A clamp will be placed on the earlobe for 60 seconds. When pain VAS of the earlobe become more than 60 mm, pain pressure threshold will be evaluated again
Fear to movement | Baseline and 48-72h post-intervention
  To assess fear to movement using the TAMPA Scale of Kinesiophobia (TSK). Scores range from 1 (totally disagree) to 4 (totally agree). The final score can range between 11 and 44 points. Higher scores indicate greater perceived fear of movement.
Catastrophizing of pain | Baseline and 48-72h post-intervention
  To assess catastrophizing of pain using the Pain Catastrophizing Scale (PCS). Scores range from 0 (nothing at all) to 4 (all the time). The final score range from 0 to 52. Higher scores indicate greater levels of catastrophism

SECONDARY OUTCOMES:
Pain intensity and interference | Baseline and 48-72h post-intervention
  To assess pain intensity and interference using the Brief Pain Inventory (BPI). Scores range from 0 (no pain/does not interfere) to 10 (worst pain imaginable/completely interferes). Higher scores indicate greater intensity and interference.
Pain vigilance and awareness | Baseline and 48-72h post-intervention
  To assess awareness, consciousness, vigilance and observation of pain using the Pain Vigilance and Awareness Questionnaire (PVAQ). Scores range from 0 (never) to 5 (always). The total scores range between 0 and 80. Higher scores indicate greater awareness, consciousness, vigilance and observation of pain.
Pain beliefs | Baseline and 48-72h post-intervention
  To assess fear and avoidance beliefs using Fear and Avoidance Beliefs Questionnaire (FABQ). Scores range from 0 (totally disagree) to 6 (totally agree). The total score range from 0 to 96. Higher scores indicate a higher degree of fear avoidance beliefs.
Health related quality of life | Baseline and 48-72h post-intervention
  To assess quality of life using the EuroQol-5D. Total score range from 1 (best health status) to 0 (death). The second part of the euroqol-5d is visual analogue scale that goes from 0 (worst state of health imaginable) to 100 (best state of health imaginable).
Pain self-efficacy | Baseline and 48-72h post-intervention
  To assess pain-self efficacy using 10 items Pain Self-Efficacy Questionnaire (10-PSEQ). Scores range from 0 (not at all confident) and 6 (completely confident). A total score range from 0 to 60. Higher scores reflect stronger self-efficacy beliefs.
Sleep quality | Baseline and 48-72h post-intervention
  To assess sleep quality using a numeric scale from 0 (worst sleep quality) to 10 (best sleep quality). Higher scores indicate greater sleep quality
Disability | Baseline and 48-72h post-intervention
  To assess disability using the Oswestry Disability Index (ODI). Total scores range from 0% (no limitation) to 100% (maximum functional limitation). Higher scores indicate higher levels of disability.
Functional status | Baseline and 48-72h post-intervention
  To assess functional status using the Patient-Specific Functioning Scale (PSFS). Scores range from 0 to 10. Higher scores indicating better functional status
Mobility | Baseline and 48-72h post-intervention
  To assess mobility using the Fingertip-to-Floor test. It will be used to examine the ability to bend forward while standing, measuring the distance between the tip of the longest finger and the floor. Lower scores are associated with decreased symptoms across all outcome measures.

OTHER OUTCOMES:
Motivation for Treatment | Baseline
  To assess motivation to treatment with the 15-item Treatment Self-Regulation Questionnaire (TSRQ). Scores range from 1 to 7 per item. Higher scores indicate greater motivation
Treatment-Generated motivation | 48-72h post-intervention
  To assess treatment-generated motivation with the 22-item Intrinsic Motivation Inventory (IMI). Scores range from 1 to 7 per item. Higher scores indicate greater motivation
Satisfaction with the intervention | 48-72h post-intervention
  To assess satisfaction with the intervention with numeric scale from 0 (no satisfaction) to 10 (completely satisfaction). Higer scores indicate higher levels of satisfaction.
Adverse events | During the intervention
  To measure the number of adverse events that may occur during the intervention.
Pain vigilance | During the intervention
  To assess pain vigilance during the intervention with a numeric scale from 0 (none) to 10 (continuously).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Granada, Granada, Spain